CLINICAL TRIAL: NCT04805320
Title: Association of Periodontal Inflammation on Immune Response in Wound Healing
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0257-21-FB
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Inflammation of Mouth
Keywords: periodontitis; wound healing; extraction
MeSH Terms: conditions — Stomatitis; Periodontitis | interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Soft tissue biopsies will be cryopreserved and prepared for ssRNA sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Dental Extraction — Extraction

SUMMARY:
Subjects who are in need of extraction of a posterior tooth will be recruited for this study. Prior to extraction, periodontal clinical markers of inflammation, body-mass index and dental radiographs will be measured/taken. The posterior tooth will be atraumatically extracted and a small soft tissue biopsy of the extraction site will be taken. At the two week follow-up, sutures will be removed and another small biopsy of soft tissue will be taken. Subjects will be seen again at 3 months for a final collection of clinical data and radiographs.

DETAILED DESCRIPTION:
Twenty-five healthy adult subjects (aged 21-70) requiring extraction of a posterior tooth will be recruited for this study. Prior to extraction, a limited-view cone beam computed tomography radiograph will be taken as well as clinical measures of periodontal inflammation (probing depths, recession, bleeding on probing, gingival crevicular fluid sampling). The extraction will be completed atraumatically and with local anesthesia. Following extraction, a small biopsy of the soft tissue of the extraction site will be taken and the site then sutured. At the two-week postoperative visit, sutures will be removed and another soft tissue biopsy of the healing site will be collected (along with clinical data from the adjacent teeth). The soft tissue biopsies will be fixed and processed for inflammatory endocytes present during wound healing. At the three-month postoperative visit, all clinical parameters of wound healing will be evaluated; including inflammatory measures (probing depths, recession, bleeding on probing, gingival crevicular fluid sampling) from the adjacent teeth; as well as a limited-view cone beam computed tomography radiograph.

The biopsies will be processed to obtain single cell counts with half of the preparation stained and analyzed via multiparameter flow cytometry. The other half of single cells obtained from the tissue biopsies will be cryopreserved for cellular indexing of transcriptomes and epitopes-sequencing.

ELIGIBILITY:
Inclusion Criteria:

* non-restorable posterior tooth (molar/premolar) in need of extraction

Exclusion Criteria:

* systemic disease that effects inflammation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults ages 21-70 with non-restorable posterior tooth requiring extraction.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cells | 3 months
  Number of inflammatory cells present

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Bavitz, DMD, Study Chair — University of Nebraska, College of Dentistry
Locations (1):
- University of Nebraska, College of Dentistry, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No